CLINICAL TRIAL: NCT00067327
Title: Treatment of Multiple Sclerosis Using Over the Counter Inosine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R21AT001301-01A1 (NIH)
Record Dates: First submitted 2003-08-15; First posted 2003-08-19 (Estimated); Last update posted 2006-03-17 (Estimated); Status verified 2006-03

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Relapsing remitting multiple sclerosis; Multiple sclerosis; Peroxynitrite; Uric acid; Inosine
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Inosine

INTERVENTIONS:
Drug: Inosine

SUMMARY:
The purpose of this study is to determine whether raising low levels of the natural antioxidant uric acid by the administration of a precursor, inosine, has any therapeutic effect on the progression of Relapsing Remitting Multiple Sclerosis (RRMS) and secondary progressive Multiple Sclerosis (MS).

DETAILED DESCRIPTION:
Uric acid is a natural inhibitor of certain chemistries associated with peroxynitrite, a product of inflammation. In animal models of multiple sclerosis (MS), these chemical reactions have been associated with breakdown of the blood-brain barrier and CNS tissue damage. In addition, MS patients have serum uric acid levels that are lower than age- and sex- matched healthy individuals. The primary purpose of this study to determine whether raising low serum uric acid levels by daily oral administration of its precursor inosine has an effect on the cumulative number of newly active lesions on magnetic resonance imaging (MRI) and to evaluate the safety and tolerability of inosine in patients diagnosed with relapsing remitting and secondary progressive MS.

ELIGIBILITY:
Inclusion Criteria:

* Nonpregnant, nonlactating females
* Females of child bearing potential must have a negative human chorionic gonadotropin (HCG) test result within 60 days before the first dose of study material.
* Males and females must practice adequate contraception, in the judgement of the investigator, during the course of the study.
* Subjects must have a diagnosis of clinically definite Relapsing Remitting Multiple Sclerosis based on medical history, physical examination, laboratory test results, and neurologic examination. Alternatively, subjects may have clinically probable MS characterized by 1 attack and the presence of at least 4 lesions on MRI within 12 months before the initial baseline evaluation.
* Subjects must have an Expanded Disability Status Scale (EDSS) test result of less than or equal to 5.0 within 60 days before the first dose of study material.
* Subjects will have serum uric acid levels less than 5 mg/dl.
* Have 1 clinical relapse in the last year

Exclusion Criteria:

* Presence of any medical disability or laboratory test result that, in the judgement of the investigator, would interfere with assessment of the tolerability, safety, or efficacy of study material or would compromise the subject's ability to provide informed consent.
* Evidence of active infection characterized by requiring treatment with antibiotics within 7 days before the first dose of study material.
* Treatment with interferons, glatiramer acetate, lymphoid irradiation, cyclophosphamide, or with other immune modifying treatments within 3 months, or corticosteroids within 1 month before the initial baseline MRI assessment in this trial.
* Recent history (within the previous 2 years) of drug or alcohol abuse.
* Known allergy to Inosine products or history of anaphylaxis.
* Previous randomization into this study.
* Treatment with an investigational agent within 30 days before the first dose of study material.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30
Dates: Start 2002-02; Study Completion 2005-09

CONTACTS AND LOCATIONS:
Overall Officials: Douglas C Hooper, PhD, Principal Investigator — Thomas Jefferson University; Hilary Koprowski, MD, Study Director — Department of Microbiology and Immunology, Thomas Jefferson University
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Hooper DC, Spitsin S, Kean RB, Champion JM, Dickson GM, Chaudhry I, Koprowski H. Uric acid, a natural scavenger of peroxynitrite, in experimental allergic encephalomyelitis and multiple sclerosis. Proc Natl Acad Sci U S A. 1998 Jan 20;95(2):675-80. doi: 10.1073/pnas.95.2.675. PMID 9435251
- [Background] Hooper DC, Scott GS, Zborek A, Mikheeva T, Kean RB, Koprowski H, Spitsin SV. Uric acid, a peroxynitrite scavenger, inhibits CNS inflammation, blood-CNS barrier permeability changes, and tissue damage in a mouse model of multiple sclerosis. FASEB J. 2000 Apr;14(5):691-8. doi: 10.1096/fasebj.14.5.691. PMID 10744626
- [Background] Koprowski H, Spitsin SV, Hooper DC. Prospects for the treatment of multiple sclerosis by raising serum levels of uric acid, a scavenger of peroxynitrite. Ann Neurol. 2001 Jan;49(1):139. doi: 10.1002/1531-8249(200101)49:13.0.co;2-a. No abstract available. PMID 11198290
- [Background] Spitsin S, Hooper DC, Leist T, Streletz LJ, Mikheeva T, Koprowskil H. Inactivation of peroxynitrite in multiple sclerosis patients after oral administration of inosine may suggest possible approaches to therapy of the disease. Mult Scler. 2001 Oct;7(5):313-9. doi: 10.1177/135245850100700507. PMID 11724447